CLINICAL TRIAL: NCT06951529
Title: The Effect of Reproductive Violence Education Given to Women on Perception of Violence, Conflict Resolution Styles and Awareness of Violence: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SBU-AYDINKARTAL-ALEYNATEZ
Record Dates: First submitted 2025-03-20; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-10

CONDITIONS: Perception of Violence; Conflict Resolution Styles
Keywords: violence; reproductive period; woman; midwifery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Intervention : control group (n:40) (No Intervention): No intervention will be made to the control group.
- Experimental : intervention group (n:40) (Experimental): In the second phase of the study, women in the intervention group will receive a 4-hour training on reproductive violence and brochures on reproductive violence will be distributed. The training will be given in the form of a powerpoint presentation and case discussion in the meeting hall of the Hamidiye Faculty of Health Sciences. Before the training, the "Informed Voluntary Consent Form", "Introductory Information Form", "Reproductive Violence Perception Form/Scale" and "Conflict and Violence Awareness Scale" will be applied to the intervention group. After the training, the "Reproductive Violence Perception Form/Scale" and "Conflict and Violence Awareness Scale" will be applied. As a follow-up test, the "Reproductive Violence Perception Form/Scale" and "Conflict and Violence Awareness Scale" will be applied after 4-6 weeks.
  Interventions: Other: Reproductive violence education

INTERVENTIONS:
Other: Reproductive violence education — The training content, which was created by obtaining expert opinions based on literature, will cover the violence that women are exposed to or may be exposed to according to the cycles they experience during their reproductive years. Definition of Violence and Its Effects on Women's Health, Adolescence and Menstruation Period Violence, Family Planning and Infertility Violence, Pregnancy and Birth-Related Violence, Menopause-Related Violence, Legal Processes in Combating Reproductive Violence.
  Arms: Experimental : intervention group (n:40)

SUMMARY:
This study was planned as a methodological and randomized controlled experimental study to determine the effects of reproductive violence education given to women on women's perceptions of violence. H0a: There is no difference in the perception levels of reproductive violence between women who were given and those who were not given reproductive violence education.

H1a: There is a difference in the perception levels of reproductive violence between women who were given and those who were not given reproductive violence education.

H0b: There is no difference in the conflict resolution styles and violence awareness levels between women who were given and those who were not given reproductive violence education.

H1b: There is a difference in the conflict resolution styles and violence awareness levels between women who were given and those who were not given reproductive violence education.

In the second phase of the study, 4 hours of reproductive violence education will be given to women in the intervention group and brochures on reproductive violence will be distributed. The education will be held in the meeting hall of Hamidiye Faculty of Health Sciences in the form of a powerpoint presentation and case discussion. Before the training, the "Informed Consent Form", "Introductory Information Form", "Reproductive Violence Perception Form/Scale" and "Conflict and Violence Awareness Scale" will be applied to the intervention group. After the training, the "Reproductive Violence Perception Form/Scale" and "Conflict and Violence Awareness Scale" will be applied. As a follow-up test, the "Reproductive Violence Perception Form/Scale" and "Conflict and Violence Awareness Scale" will be applied after 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being literate
* Being a volunteer to participate in the research
* Being a female administrative staff other than academic staff working within the Health Sciences University Hamidiye Complex

Exclusion Criteria:

* Being in menopause

  * Having a mental health problem that would prevent participation in the study
  * Receiving psychiatric treatment
  * Being an adolescent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | Baseline (10 mn)
  Women's age, socio-demographic characteristics, parameters related to violence are questioned. It will be created based on literature.
Reproductive Violence Perception Form | Baseline (10 mn)
  It includes questions about physical, psychological, economic, sexual and emotional violence during the reproductive period.
Conflict and violence awareness scale (CVV) | Baseline (10 mn)
  It was developed by the Ohio Education Commission in 2002 and its validity and reliability study was conducted by Sargin in 2010. CSFQ, which can be applied to adolescents and adults, is a five-point scale containing 27 categorical symptom items. (1. Strongly disagree, 2. Disagree, 3. Partially agree, 4. Agree, 5. Strongly agree). There is no reversed item. The high score obtained from the total of the items in the scale indicates that the individual has a high level of awareness regarding conflict and violence. The min-max score range of the CSFQ scale is 27-135. The internal consistency coefficient of the scale was found to be 0.87.

SECONDARY OUTCOMES:
Reproductive Violence Perception Form | Post-test after training (10 mn)
  It includes questions regarding physical, psychological, economic, sexual and emotional violence applied during the reproductive period.
Conflict and violence awareness scale (CVV) | Post-test after training (10 mn)
  It was developed by the Ohio Education Commission in 2002 and its validity and reliability study was conducted by Sargin in 2010. CSFQ, which can be applied to adolescents and adults, is a five-point scale containing 27 categorical symptom items. (1. Strongly disagree, 2. Disagree, 3. Partially agree, 4. Agree, 5. Strongly agree). There is no reversed item. The high score obtained from the total of the items in the scale indicates that the individual has a high level of awareness regarding conflict and violence. The min-max score range of the CSFQ scale is 27-135. The internal consistency coefficient of the scale was found to be 0.87.

OTHER OUTCOMES:
Reproductive Violence Perception Form | 4 weeks after training (10 mn)
  It includes questions regarding physical, psychological, economic, sexual and emotional violence applied during the reproductive period.
Conflict and violence awareness scale (CVV) | 4 weeks after training (10 mn)
  It was developed by the Ohio Education Commission in 2002 and its validity and reliability study was conducted by Sargin in 2010. CSFQ, which can be applied to adolescents and adults, is a five-point scale containing 27 categorical symptom items. (1. Strongly disagree, 2. Disagree, 3. Partially agree, 4. Agree, 5. Strongly agree). There is no reversed item. The high score obtained from the total of the items in the scale indicates that the individual has a high level of awareness regarding conflict and violence. The min-max score range of the CSFQ scale is 27-135. The internal consistency coefficient of the scale was found to be 0.87.

IPD SHARING:
Plan to Share IPD: Yes